CLINICAL TRIAL: NCT05837663
Title: Trifecta-Lung cfDNA-MMDx Study: Comparing the Dd-cfDNA Test to MMDx Microarray Test and Central HLA Antibody Test
Brief Title: Trifecta-Lung cfDNA-MMDx Study
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Natera, Inc. (Industry); One Lambda (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00048176
Record Dates: First submitted 2023-04-03; First posted 2023-05-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplantation
Keywords: Donor derived cfDNA; Gene expression; Lung transplant biopsy; Blood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA isolated from patient biopsy cfDNA isolated from patient blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Demonstrate the relationship between dd-cfDNA levels and HLA antibodies in blood transplant recipient and Demonstrate the Molecular Microscope® (MMDx) Diagnostic System results in indication and protocol biopsies from lung transplants.

DETAILED DESCRIPTION:
The current standard for assessment of rejection in lung transplants is a transbronchial biopsy (TBB) interpreted by histology according to International Society of Heart and Lung Transplantation (ISHLT) guidelines. This has considerable error rates, many due to the high disagreement among pathologists. There is a need for new methods of assessing TBBs. Furthermore, by analyzing different types of biopsies (TBBs and endobronchial - 3BMBs), we hope to improve the safety of the biopsy procedure, while maintaining its accuracy. The emergence of blood donor-derived cell-free DNA (dd-cfDNA) measurement offers a new opportunity for screening for rejection. To address the unmet need for precision and accuracy, the Alberta Transplant Applied Genomics Centre (ATAGC, University of Alberta) has developed a new diagnostic system - the Molecular Microscope® Diagnostic System (MMDx), which uses microarrays to define the genome-wide gene expression and interpret lung transplant rejection and injury ((chronic lung allograft dysfunction (CLAD) related changes)). Now a new screening test is being introduced: the monitoring of dd-cfDNA released in the blood by the heart during rejection. The Natera Inc dd-cfDNA Prospera® test is based on the massively multiplex polymerase chain reaction that targets 13,392 single nucleotide polymorphisms and targeted sequences are quantified by Next Generation Sequencing. The Prospera® test has been done on kidney transplant recipients and detected "active rejection" and differentiated it from borderline rejection and no rejection. However, Prospera® test was not examined (the dd-cfDNA results) in lung transplant recipients. dd-cf-DNA test for lung transplants must now be calibrated against MMDx that is based on global gene expression, the new standard for biopsy interpretation. The present study will calibrate centrally measured (Natera Inc) dd-cfDNA levels obtained at the time of an indication or protocol biopsy against the MMDx measurements of T cell-mediated rejection (TCMR), antibody-mediated rejection (ABMR-like) and tissue injury. The present study will compare dd-cfDNA and MMDx in 600 prospectively collected TBBs and 3BMBs for clinical indications and protocol, and accompanying 1800 blood samples, to calibrate the dd-cfDNA (Natera Inc.) levels against the MMDx biopsy diagnoses of TCMR, ABMR-like (and its stages), and injury, as well as central assessment of Human Leukocyte Antibody (HLA) antibody (One Lambda), interpreted centrally as donor specific antibody (DSA) based on the tissue typing results. This study is an extension of the INTERLUNG ClinicalTrials.gov identifier: NCT02812290.

Currently the study accrued 108 paired TBBs and 3BMBs, 9 TBBs, and 64 corresponding blood samples for dd-cfDNA test.

ELIGIBILITY:
Inclusion Criteria:

Adult, Older adult

Exclusion Criteria:

Patients will be excluded from the study if they decline participation Are unable to give informed consent. Recipients of multiple organs, cancer patients and pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult lung transplant recipients undergoing indication biopsy for suspected graft dysfunction will be eligible.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Calibration of Prospera® test for T cell mediated rejection | 18 months
  Set dd-cfDNA test cut-off values against the probability of T cell-mediated rejection in the biopsy (TBB and 3BMB) as reported by MMDx. Calibration of dd-cfDNA test cut-off values against the probability of T cell-mediated rejection in the biopsy as reported by MMDx.
Calibration of Prospera® test for antibody-mediated rejection | 18 months
  Set dd-cfDNA test cut-off values against the probability of antibody-mediated rejection in the biopsy (TBB and 3BMB) as reported by MMDx.
Calibration of Prospera® test for lung injury | 18 months
  Set dd-cfDNA test cut-off values against the probability of acute and chronic lung injury in the biopsy (TBB and 3BMB)as reported by MMDx.
Report calibrated Prospera® test results for rejection | 6 months
  Report new dd-cfDNA test cut-off values for rejection
Report calibrated Prospera® test results for lung injury | 6 months
  Report new DD-cfDNA test cut-off values for lung injury

SECONDARY OUTCOMES:
Assessment of donor-specific antibody status | 6 months
  Record and compare the DSA status (positive or negative) based on centralized and local HLA antibody to histology diagnoses..
.Estimate the false positive rate of dd-cfDNA for MMDx and histology in indication and protocol biopsies | 6 months
  Calculate the sensitivity and specificity of dd-cfDNA for MMDx and histology diagnoses.
Determine whether calibrated dd-cfDNA blood test will replace biopsies | 6 months
  Determine if dd-cfDNA test will avoid need for indication biopsy when transplant function deteriorates - yes or no. This will be based on the consensus between participating clinicians.
Determine whether calibrated dd-cfDNA blood test predicts the effect of treatment | 6 months
  Determine the values for dd-cfDNA for grades of response to treatment: no change, partial response, complete resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD PhD, Principal Investigator — Alberta Transplant Applied Genomics Centre, University of Alberta
Locations (18):
- United States (11):
  - St. Joseph's Hospital and Medical Center 350 West Thomas Road, Floor 8HLT, Phoenix, Arizona
  - Division of Pulmonary, Critical Care and Sleep Medicine, University of Florida, College of Medicine, Gainesville, Florida
  - USF Health, Morsani College of Medicine, 12901 Bruce B. Downs Blvd. MDC40, Tampa, Florida
  - Indiana University Methodist Hospital 1812 N. Capitol Ave Suite W131L, Indianapolis, Indiana
  - Johns Hopkins Interventional Pulmonology, Sheikh Zayed Tower, Room 7125L, 1800 Orleans Street, Baltimore, Maryland
  - Division of Pulmonary, Allergy & Critical Care Medicine Columbia University Irving Medical Center, New York, New York
  - The Ohio State University Wexner Medical Center, 410 W 10th Ave, Columbus, Ohio
  - BAYLOR SCOTT & WHITE RESEARCH INSTITUTE , 3409 Worth Street, Dallas, Texas
  - UT Southwestern Medical Center, 5939 Harry Hines Blvd., Dallas, Texas
  - Houston Methodist Lung Transplant Center, 6550 Fannin St., SM1001, Houston, Texas
  - UT Health San Antonio 7703 Floyd Curl Drive, MSC: 7858, San Antonio, Texas
- The Alfred Hospital, Monash University, Melbourne, Australia
- Department of Thoracic Surgery, Medical University of Vienna, Vienna, Austria
- Canada (3):
  - Department of Medicine, University of Alberta, Edmonton, Alberta
  - Alberta Transplant Applied Genomics Centre, University of Alberta, Edmonton, Alberta
  - University Health Network, Toronto General Hospital, Toronto, Ontario
- Czechia (2):
  - Motol University Hospital, V Uvalu 84, Prague
  - Charles University/Hospital Motol, Prague

IPD SHARING:
Plan to Share IPD: No
Only IPD data will be shared within a participating center